CLINICAL TRIAL: NCT05361434
Title: A Prospective Observational International Study of Cabozantinib Tablets in Combination With Nivolumab as First-line Treatment of Advanced Renal Cell Carcinoma in Adults
Brief Title: A Study of the Effectiveness of Cabozantinib in Combination With Nivolumab as First-line Treatment of Advanced Renal Cell Carcinoma (aRCC) in Adults
Acronym: CaboCombo
Status: Active, not recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60000-452
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect data to describe the safety and effectiveness of cabozantinib and nivolumab in combination as a first-line treatment in adults with aRCC with clear cell-component, according to real-world clinical practice. The decision to prescribe cabozantinib and nivolumab in combination will be made prior to, and independently from, the decision to enrol the participant in study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of aRCC with clear-cell component
* Participants with no prior systemic treatment for aRCC with clear-cell component;
* Physician-initiated decision to treat with cabozantinib and nivolumab in combination (prior to study enrolment), according to Cabometyx® and Opdivo® approved local labels;

Exclusion Criteria:

* Current participation in an investigational program with any intervention which could possibly interfere the treatment and impact this study;
* History of allergy or hypersensitivity to Cabometyx® or Opdivo® components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include participants with advanced renal cell carcinoma with clear cell component, for whom a decision to treat with cabozantinib and nivolumab in combination has been made by the treating physician
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) rate (death of any cause) from the start of cabozantinib in combination with nivolumab. | At 18 months follow up

SECONDARY OUTCOMES:
Tumor median progression-free survival (PFS) time | Every month until month 4, and every 3 months after month 4 up to 42 month or disease progression
  Including clinical and radiographic assessments defined as the time between the start date of cabozantinib in combination with nivolumab and the date of progression or death of any cause. The Kaplan-Meier method will be used to estimate median PFS.
Proportion of participants who achieve partial or complete response (Objective Response Rate (ORR)) | Every month until month 4, and every 3 months after month 4 up to 42 month or disease progression
  Assessed by the investigator
Duration of response (DOR) | Every month until month 4, and every 3 months after month 4 up to 42 month or disease progression
  Defined as the interval from the date of first response (complete or partial) to treatment with cabozantinib in combination with nivolumab, to progressive disease or death
Proportion of participants who achieve complete response, partial response or stable disease (Disease Control Rate (DCR)). | Every month until month 4, and every 3 months after month 4 up to 42 months or disease progression.
Time of response (TTR) | Every month until month 4, and every 3 months after month 4 up to 42 months or disease progression
  Defined as the time between the start date of cabozantinib in combination with nivolumab and date of first response (complete or partial).
Pattern of use of cabozantinib under real-world practice conditions. | Every month until month 4, and every 3 months after month 4 up to 42 months or disease progression
Pattern of use of nivolumab under real-world practice conditions. | Every month until month 4, and every 3 months after month 4 up to 42 months or disease progression
Incidence of treatment-emergent Adverse Events (TEAEs) including nonserious Adverse Events (AEs), and Serious Advers Events (SAEs). | Up to 42 months or disease progression
  All AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) and will be classified by MedDRA PT and SOC.
Change in disease-related symptoms | Change from baseline at each visit up to 42 months
  Assessed by the Functional Assessment of Cancer Therapy Kidney Cancer Symptom Index - Disease Related Symptoms (FKSI-DRS) questionnaire
Change in pain | Change from baseline at each visit up to 42 months
  Assessed by the Numerical Pain Rating Scale (NPRS)
Percentage of participants receiving subsequent anticancer therapies following cabozantinib and nivolumab discontinuation | Up to 42 months.
  Including: Sequences of treatment; drug names and duration of treatment; and reason for end of treatment line

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (66):
- Belgium (3):
  - CHU St Pierre & Brugmann, Brussels
  - Jessa Ziekenhuis, Hasselt
  - CHU Namur Mont-Godinne, Yvoir
- France (39):
  - Centre Hospitalier Universitaire (CHU) de Angers, Angers
  - Hopital de Mercy- CHR Metz Thionville, Ars-Laquenexy
  - Institut Ste Catherine - Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier Régional Universitaire de Besançon - Jean Minjoz, Besançon
  - ICONE, Bezannes
  - Groupe Hospitalier Saint-André (Bordeaux), Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier de Boulogne-sur-mer, Boulogne-sur-Mer
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Centre Finisterien de Radiotherapie et d'Oncologie, Brest
  - Centre d'Urologie Site Médipole - Centre Catalan d'Urologie, Cabestany
  - Centre de Lutte Contre le Cancer Jean PERRIN, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire (CHU) Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Institut de Cancérologie de Bourgogne, Dijon
  - Centre Hospitalier Annecy Genevois, Épagny
  - Centre Hospitalier intercommunal Saint Raphaël Frejus, Fréjus
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Groupe Hospitalier De La Rochelle - Ré - Aunis, La Rochelle
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Hôpital Privé Le Bois, Lille
  - Hopital Privé Jean Mermoz, Lyon
  - Centre Hospitalier Universitaire (CHU) de Nantes - Hôtel-Dieu, Nantes
  - Centre Hospitalier Régional D'orléans, Orléans
  - Centre Hospitalier Tenon, Paris
  - Hopital Bichat -Claud Bernard, Paris
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers
  - CHU Charles Nicolle, Rouen
  - Clinique Mathilde Oncologie médicale, Rouen
  - Centre d'Oncologie de l'Estuaire, Saint-Nazaire
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hospital Foch - Oncology Service, Suresnes
  - Hospital Foch - Urology Service, Suresnes
  - Centre Hospitalier Régional Universitaire de (CHRU) de Tours - Hôpital Bretonneau, Tours
  - CH Dentellières, Valenciennes
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
- Greece (4):
  - General Hospital of Athens Alexandra, Athens
  - Henry Dunant Hospital, Athens
  - ATTIKO University Hospital, Chaïdári
  - Papageorgiou General Hosp of Thessaloniki, Thessaloniki
- Italy (11):
  - Ospedale Generale Provincial, Macerata
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", IRCCS - Oncologia, Meldola
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - AOU San Luigi Gonzaga, Orbassano
  - IOV - Istituto Oncologico Veneto - IRCCS - Ospedale Busonera, Padua
  - P.O Santa Maria delle Grazie, ASL Napoli 2 Nord, Pozzuoli
  - Ospedale "Santa Maria delle Croci" di Ravenna, Ravenna
  - Ospedale San Camillo Forlanini, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - PU A.Gemelli, Università Cattolica del Sacro Cuore, Roma
- Akershus Universitetssykehus, Lørenskog, Norway
- Saudi Arabia (2):
  - King Abdulaziz Medical City - Jeddah, Jeddah
  - King Abdulaziz Medical City- Riyadh, Riyadh
- South Korea (4):
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- United Kingdom (2):
  - Belfast City Hospital, Belfast
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Barthelemy P, Dutailly P, Qvick B, Perrot V, Verzoni E. CaboCombo: a prospective, phase IV study of first-line cabozantinib + nivolumab for advanced renal cell carcinoma. Future Oncol. 2024 Apr;20(13):811-819. doi: 10.2217/fon-2023-0353. Epub 2023 Jul 5. PMID 37403652